CLINICAL TRIAL: NCT05054218
Title: Immunogenicity of a Third Dose of mRNA-1273 Vaccine (Moderna) Among Cancer Patients
Brief Title: COVID-19 Immunogenicity of a Third Dose of mRNA-1273 Vaccine Among Cancer Patients
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MCC-21536
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Covid19; SARS-CoV2 Infection
Keywords: Immunogenicity; Antibodies; Vaccine Adverse Events
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Draw: One (1) 10 ml tiger-top tube Blood Draw: Two (2) 8 ml CPT tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participants who receive 3rd dose of mRNA-1273 SARS-CoV-2 vaccine: Cancer patients who have already received their 1st and 2nd doses of mRNA-1273 SARS-CoV-2 vaccine will receive a 3rd dose of the vaccine. The volume of vaccine injected will be 0.5 mL, containing a 100-μg dose of mRNA-1273.
  Interventions: Biological: mRNA-1273

INTERVENTIONS:
Biological: mRNA-1273 — Participants will receive a 0.5 mL injection of the vaccine that contains a 100-μg dose of mRNA1273. The vaccine will be administered into the deltoid muscle.

SUMMARY:
Investigators will evaluate the immunogenicity of a third dose of mRNA-1273 SARS-CoV-2 vaccine among cancer patients receiving the recommended third vaccine dose

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Is a cancer patient enrolled in the Cancer Patient Immune Response to COVID-19 Vaccine study (a basic science study) MCC 21138 or who has completed the two mRNA-1273 vaccine series prior to March 31, 2021.
* Understands, agrees and is able to comply with the study procedures and provides written informed consent.
* Has no known or suspected allergy or history of anaphylaxis, urticaria, or other significant adverse reactions to the vaccine or its excipients.
* Has not received more or less than 2 doses of mRNA-1273 vaccine

Exclusion Criteria:

* Participants who will not return for the third vaccine dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Moffitt Cancer Center who have completed their two-dose series of the mRNA-1273 vaccine prior to March 31, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-07-16 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
1. The level of anti-SARS-CoV-2 Spike (S)-specific neutralizing antibody (nAb) 28 days post-dose 3 | 28 days
  The level of anti-SARS-CoV-2 Spike (S)-specific neutralizing antibody (nAb) up to study day 28 will be measured by specific neutralizing antibody and serum assays
Anti-SARS-CoV-2 Spike (S)-specific neutralizing antibody (nAb) 6 months post-dose 3 | 6 months
  The level of anti-SARS-CoV-2 Spike (S)-specific neutralizing antibody (nAb) up to study month 6 will be measured by specific neutralizing antibody and serum assays
Anti-SARS-CoV-2 Spike (S)-GMT Ab 28 days post-dose 3 | 28 days
  The level of anti-SARS-CoV-2 Spike (S)-GMT Ab up to study day 28 will be measured by specific neutralizing antibody and serum assays
Anti-SARS-CoV-2 Spike (S)-GMT Ab 6 months post-dose 3 | 6 months
  The level of anti-SARS-CoV-2 Spike (S)-GMT Ab up to study month 6 will be measured by specific neutralizing antibody and serum assays
Level antibodies that block the binding of ACE2 to RBD antigens from 10 SARS-CoV-2 variants of concern 28 days post-dose 3 | 28 days
  The level antibodies that block the binding of ACE2 to RBD antigens from 10 SARS-CoV-2 variants of concern up to study day 28 will be measured by specific neutralizing antibody and serum assays
Level antibodies that block the binding of ACE2 to RBD antigens from 10 SARS-CoV-2 variants of concern 6 months post-dose 3 | 6 months
  The level antibodies that block the binding of ACE2 to RBD antigens from 10 SARS-CoV-2 variants of concern up to study month 6 will be measured by specific neutralizing antibody and serum assays

SECONDARY OUTCOMES:
Solicited local and systemic adverse reactions (ARs) post-dose 3 up to study day 20 | Up to 20 days
  Investigators will measure solicited local and systemic adverse reactions (ARs) at day 14 (+/- 5 days) post 3rd dose of vaccine
Solicited local and systemic adverse reactions (ARs) post-dose 3 up to study day 40 | Up to 42 days
  Investigators will measure solicited local and systemic adverse reactions (ARs) at day 28 (+ 14 days) post 3rd dose of vaccine
Number of participants who experienced Serious Adverse Events and Adverse Events | Baseline thru up to 6 months
  Participants able to safely tolerate a 3rd dose of mRNA-1273 vaccine as measured by adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Giuliano, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinical-trials-research/clinical-trials/